CLINICAL TRIAL: NCT04923295
Title: The Effect of Dapagliflozin on Ultrafiltration Among Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: An-Najah National University (Other)
Responsible Party: Principal Investigator, Zakaria Hamdan, Assistant Professor of Medicine, An-Najah National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2 PD
Record Dates: First submitted 2021-05-25; First posted 2021-06-11 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Peritoneal Dialysis Complication; Ultrafiltration Failure
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Pre and post intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre Treatment and post treatment (Experimental): Patients on Peritoneal Dialysis will be evaluated by PET and transport status Patients on Peritoneal Dialysis will be evaluated by PET after treatment with Dapagliflozin
  Interventions: Drug: Dapagliflozin 10Mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Effect of Dapagliflozin on ultrafiltration and PET results among peritoneal dialysis patients
  Other Names: Forxiga 10mgs

SUMMARY:
Patients with average or high average peritoneal glucose transport status be included in the study as mentioned in the inclusion and exclusion criteria.

The change in peritoneal glucose transport will be evaluated before and after one month treatment with 10 mg of Dapagliflozin.

Peritoneal Equilibration Test (PET) test for patients before and after Dapagliflozin use and volume status of patients as measured by ultrafiltration from peritoneal dialysis exchanges.

The aim of the trial is to determine whether dapagliflozin can decrease glucose absorption from peritoneal fluid and reduce plasma glucose absorption from the PD fluid and thus improve ultrafiltration with a reduction in intraperitoneal glucose exposure

DETAILED DESCRIPTION:
The research targets patients on peritoneal dialysis with average and high transport status documented by Peritoneal Equilibrium Transport Test (PET test) in Najah National University Hospital.

Research participants will be recruited from the patients on peritoneal dialysis in NNUH. A study team member will prescreen the patient based upon the inclusion/exclusion criteria. If potentially eligible, the coordinator will approach candidates directly to provide information about the study and to invite them to voluntarily participate. The primary investigator will provide the participant with the informed consent document to read to read and to sign it if they agree to participate. The study includes patients on peritoneal dialysis with average and high transport status documented by Peritoneal Equilibrium Transport Test (PET test).

Prior to starting treatment with Dapagliflozin all patients included in the study population will have the following tests performed:

Modified Peritoneal Equilibrium Test with 4.5% Dextrose peritoneal fluid Hemoglobin A1C levels 24 urine collection for protein, glucose, and creatine clearance Peritoneal fluid albumin levels Patients will report daily ultrafiltration volumes one week prior to the start of treatment Blood pressure, heart rate and weight of patients prior to the start of treatment Sodium sieving will estimated by subtracting the sodium dialysate concentration at time zero from the sodium dialysate concentration at one hour. Uric Acid levels

Patients will then start on Dapagliflozin 10 mg daily for 4 weeks. During the study period patients will be evaluated for any side effects including;

Volume Depletion Ketoacidosis Hypoglycemia Urinary Tract infections Uric Acid levels Discontinuation of drug due to Adverse Events (DAEs) Changes in clinical chemistry/hematology parameters Adverse events of interest (volume depletion, major hypoglycemic events, fractures, diabetic ketoacidosis, genital and urinary tract infections)

Patients will monitored for the following:

Glucose levels Bicarbonate levels Blood pressure readings Hemoglobin A1C levels every 4 months.

Depending on the volume of ultrafiltration per patient and patient's weight, the investigators will have the choice to change the prescription; as per the investigator clinical judgment. For example if a patient with a four PD exchanges using 2.5% dextrose which yielded about 1.5L of ultrafiltration daily, and once started on Dapagliflozin had an increase ultrafiltration of 2.3 L a day, the investigator will be able to adjust the prescription to include 1.5% exchanges; resulting in less ultrafiltration volume.

At the end of the study period patient will be evaluated for the following:

Modified Peritoneal Equilibrium Test with 4.5% Dextrose peritoneal fluid 24 urine collection for protein, glucose, and creatine clearance Peritoneal fluid albumin levels Blood pressure, heart rate and weight of patients prior to the start of treatment Sodium sieving will estimated by subtracting the sodium dialysate concentration at time zero from the sodium dialysate concentration at one hour. Uric acid levels The collection of all blood pressure, hear rate reading and weights of patients will be recorded along with a daily ultrafiltration volume.

Samples of serum and peritoneal fluid effluent will be frozen -20C for any future studies.

ELIGIBILITY:
Inclusion Criteria:

* The research targets patients on peritoneal dialysis with average and high transport status documented by Peritoneal Equilibrium Transport Test (PET test) in Najah National University Hospital.

Exclusion Criteria:

1. Patients less than 18 years
2. An episode of Peritonitis in less than three months
3. History of recurrent hypoglycemia ( more than two episodes during one month prior to enrollment in the study)
4. Liver disease: Hepatic impairment aspartate transaminase [AST] or alanine transaminase [ALT] >3x the upper limit of normal [ULN]; or total bilirubin >2x ULN at time of enrolment)
5. Any allergic reaction to dapagliflozin
6. Type I DM
7. Pregnancy or women who are breast-feeding
8. Symptomatic hypotension or a mean arterial pressure (MAP) less than 60 mmHg
9. MI, unstable angina, stroke, or transient ischemic attack (TIA) within 12 weeks before enrolment
10. Active malignancy requiring treatment at the time of visit -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Mean Peritoneal Fluid Glucose ratio (D4/D0) after 4 Weeks of Treatment with 10 mg of Dapagliflozin | 4 weeks
  The mean glucose concentrations will be evaluated by the modified Peritoneal Equilibrium Test from Baseline and after 4 weeks with Dapagliflozin treatment. The modified peritoneal equilibration test (PET) characterizes the peritoneal transport of fluid, creatinine and urea using a 4.5% dextrose peritoneal fluid.The concentration of glucose in the dialysis fluid (D4) at 4 hours is divided by the glucose in the dialysis fluid at the beginning (D0), generating the D4/D0.
Change from Baseline in the Mean Ultrafiltration Volume after 4 Weeks of Treatment with 10 mg of Dapagliflozin | 4 weeks
  Ultrafiltration volume from Baseline and after 4 weeks with Dapagliflozin treatment assessment by the modified Peritoneal Equilibrium Test. The modified peritoneal equilibration test (PET) characterizes the peritoneal transport of fluid, creatinine and urea using a 4.5% dextrose peritoneal fluid.
Change from Baseline in the Mean 4 Hour Peritoneal Fluid to Plasma Creatinine (D/P) after 4 Weeks of Treatment with 10 mg of Dapagliflozin | 4 weeks
  Peritoneal Solute Transport Rate is measured with 5% or greater reduction in PSTR as measured by the modified Peritoneal Equilibrium Test. The modified peritoneal equilibration test (PET) characterizes the peritoneal transport of fluid, creatinine and urea using a 4.5% dextrose peritoneal fluid.The concentration of creatinine in the dialysis fluid (D) at 4 hours is divided by the plasma creatinine (P), generating the D/P creatinine.
Change in Peritoneal Fluid Sodium Dip 4 Weeks of Treatment with 10 mg of Dapagliflozin | 4 weeks
  Peritoneal Fluid sodium dip is done by measuring the peritoneal fluid sodium concentration at the time of infusion to the patient and after one hour of dwell time in the peritoneum.

SECONDARY OUTCOMES:
Response rate - 25 percent increase in the sodium dip at 60 minutes | 4 weeks
  The response rate was defined as the number of participants with a 25% or greater increase in in the sodium dip at 60 minutes from baseline and after 4 weeks of treatment with 10 mg of Dapagliflozin
Response rate - 25 percent increase in peritoneal fluid glucose D4/D0 | 4 weeks
  The response rate was defined as the number of participants with a 25% or greater increase in D4/D0 peritoneal fluid glucose concentration from baseline and after 4 weeks of treatment with 10 mg of Dapagliflozin
Response rate - 10 percent or greater decrease in the mean 4 hour peritoneal fluid to plasma creatinine (D/P) | 4 weeks
  The response rate was defined as the number of participants with a 10% or greater decrease in D4/D0 peritoneal fluid glucose concentration from baseline and after 4 weeks of treatment with 10 mg of Dapagliflozin
Response rate - 25 percent increase in ultrafiltration volume | 4 weeks
  The response rate was defined as the number of participants with a 25% or greater increase in ultrafiltration volume from baseline and after 4 weeks of treatment with 10 mg of Dapagliflozin
Number of Participants With Treatment-Related Adverse Events as Assessed by (CTCAE v4.0) Common Terminology Criteria for Adverse Events Version 4.0 | 6 weeks
  The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

CONTACTS AND LOCATIONS:
Overall Officials: Zakaria I Hamdan, MD, Principal Investigator — An Najah National University Hospital
Locations (1):
- An Najah National University Hospital, Nablus, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 4 weeks

REFERENCES:
- [Derived] Hamdan Z, Abdel-Hafez Y, Enaya A, Sarsour A, Kharraz L, Nazzal Z. Dapagliflozin in peritoneal dialysis patients: a pilot study evaluating peritoneal membrane function. BMC Nephrol. 2024 Jan 26;25(1):37. doi: 10.1186/s12882-023-03429-2. PMID 38279109